CLINICAL TRIAL: NCT01851902
Title: PREdicting Determinants of Atrial Fibrillation or Flutter for Therapy Elucidation in Patients at Risk for Thromboembolic Events (PREDATE AF)"
Brief Title: PREdicting Atrial Fibrillation or Flutter
Acronym: PREDATE-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Keesler Air Force Base Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FKE20130012H
Record Dates: First submitted 2013-05-02; First posted 2013-05-13 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CHA2DS2-VASc Score 2 - 4: Physicians estimate the risk of stroke in AF patients using either the CHADS2 or CHA2DS2-VASc scoring; this is a low risk cohort.
- CHA2DS2-VASc Score 5 - 6: Physicians estimate the risk of stroke in AF patients using either the CHADS2 or CHA2DS2-VASc scoring; this is a medium risk cohort.
- CHA2DS2-VASc Score 7 - 9: Physicians estimate the risk of stroke in AF patients using either the CHADS2 or CHA2DS2-VASc scoring; this is a high risk cohort.

SUMMARY:
The purpose of this study is to determine, through continuous monitoring with a cardiac monitoring device placed under the skin, the incidence of atrial fibrillation or flutter (AF). The cardiac monitor will be placed in patients without symptoms but at risk for AF. It is hoped that this information may assist health care professionals in treatment decisions related to the early identification of patients at high risk for AF.

DETAILED DESCRIPTION:
Background: Atrial fibrillation and atrial flutter (AF) are common cardiac arrhythmias that confer a substantial stroke burden largely because the vast majority of AF is asymptomatic and identified after a stroke has occurred. Until recently, only intermittent cardiac monitors were available, with most AF episodes remaining undetected due to poor sensitivity. Health care providers estimate the risk of stroke in AF patients using a patient's comorbidity profile to determine who should be treated with oral anticoagulant therapy for stroke prevention. The incidence of AF in patients with high stroke risk comorbidities is not known. The Medtronic Reveal insertable cardiac monitor (ICM) is a continuous monitoring device with excellent AF detection.

Purpose and Study Objectives: The purpose of the PREDATE AF study is to determine the incidence of AF in asymptomatic patients at high risk for having AF in order to determine which patient characteristics are most predictive of the development of AF. The primary objective is to determine the AF incidence rate; secondary objectives include identifying the most important predictors of AF onset and identifying how physicians respond once AF has been discovered.

Study Design: The trial is a prospective, single arm, open-label, single center clinical study which will enroll up to 360 patients at high risk of having AF based upon their comorbidity profile, who will then receive an ICM. Enrolled subjects will be followed for a minimum of 18 months to monitor for the detection of AF. Monthly ICM data transmissions will be the mechanism of AF detection, and this information will be utilized to determine the AF incidence rate

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the approved FDA indication to receive the ICM
* Patient is suspected, based on demographics, to be at high risk of having AF, as determined by the clinical investigator
* Patient has a CHA2DS2-VASc score ≥ 2 [Note: stroke/TIA criterion as part of the CHA2DS2-VASc score for this trial is limited to either an ischemic stroke or TIA, which occurred more than one year prior to enrollment.]
* Patient is 18 years of age or older
* Patient has a life expectancy of 18 months or more

Exclusion Criteria:

* Patient has a documented history of AF or atrial flutter
* Patient has a symptom complex consistent with an arrhythmia (where an ICM may have an alternate indication for use)
* Patient had an ischemic stroke or TIA within past year prior to enrollment
* Patient has a history of a hemorrhagic stroke
* Patient is currently implanted with a permanent pacemaker, insertable loop recorder, implantable defibrillator, cardiac resynchronization therapy device (pacemaker or defibrillator)
* NYHA Class IV Heart Failure patient
* Patient had heart surgery within previous 90 days prior to enrollment
* Patient had an MI within the previous 90 days prior to enrollment
* Patient is taking chronic immunosuppressant therapy
* Patient is taking an anti-arrhythmic drug
* Patient is contraindicated for long term anticoagulation medication
* Patient is taking a long-term anticoagulation medication
* Any concomitant condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse, emotional / psychological diagnosis)
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from the principal investigator
* Patient has a creatinine clearance <30 ml/min or is on dialysis
* Active pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The PREDATE AF trial is a prospective, single arm, open-label, single center clinical study to evaluate the incidence of AF in patients that are suspected to be at high risk of having AF, as defined by a modified CHA2DS2-VASc score.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Atrial Fibrillation | 2 years
  Incidence rate of AF calculated in each arm as the number of participants with an initial episode of AF lasting greater than or equal to six minutes divided by the total number of participants in that arm.

CONTACTS AND LOCATIONS:
Overall Officials: Javed M Nasir, MD, Study Director — Keesler Medical Center
Locations (1):
- Keesler Medical Center, Keesler Air Force Base, Mississippi, United States